CLINICAL TRIAL: NCT00782067
Title: A Single Arm, Phase II, Open-Label Study to Determine the Efficacy of 100mg Twice Daily Oral Dosing of Midostaurin Administered to Patients With Aggressive Systemic Mastocytosis or Mast Cell Leukemia +/- an Associated Hematological Clonal Non-Mast Cell Lineage Disease
Brief Title: Efficacy and Safety of Midostaurin in Patients With Aggressive Systemic Mastocytosis or Mast Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPKC412D2201; 2008-000280-42 (EudraCT Number)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Leukemia
Keywords: Aggressive systemic mastocytosis; mast cell leukemia; C-Findings; tyrosine kinase inhibitor; KIT mutation; AHNMD; Systemic; Aggressive
MeSH Terms: conditions — Leukemia; Mastocytosis, Systemic; Leukemia, Mast-Cell; Aggression | interventions — midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midostaurin (PKC412) (Experimental): Midostaurin was administered at a dose of 100 mg twice daily (bid) in continuous cycles of 28 days until disease progression, intolerable toxicity or withdrawal due to any cause, whichever occurred first.
  Interventions: Drug: Midostaurin (PKC412)

INTERVENTIONS:
Drug: Midostaurin (PKC412) — Midostaurin was provided as 25 mg soft gelatin capsules for oral administration.

SUMMARY:
The purpose of this study was to determine the efficacy and safety of twice daily (bid) oral midostaurin in patients with Aggressive Systemic Mastocytosis (ASM) or Mast Cell Leukemia (MCL) with or without an Associated Hematological clonal Non-Mast cell lineage Disease (AHNMD).

ELIGIBILITY:
Key inclusion criteria:

* Patients ≥ 18 years of age who provided written informed consent, Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 and a life expectancy of >12 weeks, electrocardiogram with a QTcF of ≤ 450 ms, with a diagnosis of SM and sub-variants based on WHO criteria.
* Patients with ASM or MCL were to have one or more measurable clinical findings (termed "C-findings") and defined as those attributable to the mast cell disease component and not to AHNMD or any other cause.
* Patients with MCL were to have BM aspirate smears with ≥ 20% immature MCs. Patients with AHNMD were eligible if it was not life-threatening or in an acute stage.

Key exclusion criteria:

* Patients with cardiovascular disease including congestive heart failure class III or IV according to the New York Heart Association classification, left ventricular ejection fraction (LVEF) of <50%, myocardial infarction within the previous 6 months, or poorly controlled hypertension.
* Patients with a heart block of any degree at screening (for Canada only).
* Patients with an AHNMD who required immediate cytoreductive therapy or targeted therapy (other than midostaurin).
* Patients who had demonstrated relapse after 3 or more prior regimens of SM treatment regardless of treatment regimen for supportive care (e.g., symptom-limiting therapies).
* Patients who had received any investigational agent, targeted therapy, chemotherapy, interferon-α, or 2 chlorodeoxyadenosine within 30 days prior to start of midostaurin treatment.
* Patients who had ASM with eosinophilia and known positivity for the FIP1L1- PDGFRα fusion unless they had demonstrated relapse or disease progression on prior imatinib therapy.
* Patients who had received any treatment with midostaurin prior to study entry.
* Patients who had received hematopoietic growth factor support within 14 days of Day 1 of midostaurin treatment.
* Patients who had any surgical procedure, excluding central venous catheter placement or other minor procedures (e.g. skin biopsy) within 14 days of Day 1 of midostaurin treatment.
* Patients with any pulmonary infiltrate, including those suspected to be of infectious origin. In particular, patients with resolution of clinical symptoms of pulmonary infection but with residual pulmonary infiltrates on chest x-ray were not eligible until the pulmonary infiltrates had completely resolved. Exception: patients with ASM/MCL ± AHNMD-related pleural effusion as judged by the Investigator and approved by the SSC Chairperson or designee were permitted to enter the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-10-13 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- United States (9):
  - University of California at Los Angeles Dept. of Hematology Clinic, Los Angeles, California
  - Stanford University Medical Center Stanford University 2, Stanford, California
  - Georgia Health Sciences University Dept.ofMedicalCollegeOfGeorgia, Augusta, Georgia
  - Dana Farber Cancer Institute Hematology / Oncology, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center DeptofMichiganCancerCenter(3), Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center Dept. of MSKCC (2), New York, New York
  - Oregon Health and Science University Dept. Hematologic Malignancies, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University SC, Richmond, Virginia
- Australia (2):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Prahran, Victoria
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Leuven, Belgium
- Canada (2):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- France (2):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Paris
- Germany (5):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
- Novartis Investigative Site, Groningen, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Gdansk, Poland
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow - Scotland
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Medawar G, Sakalabaktula K, Magri J, Rinker E, Baratam P. KIT V560D-Mutated Systemic Mastocytosis Associated With High-Risk Myelodysplastic Syndrome: A Unique Case of Systemic Mastocytosis-Associated Hematologic Neoplasm. Case Rep Hematol. 2024 Nov 30;2024:4360304. doi: 10.1155/crh/4360304. eCollection 2024. PMID 39649724
- [Derived] Hartmann K, Gotlib J, Akin C, Hermine O, Awan FT, Hexner E, Mauro MJ, Menssen HD, Redhu S, Knoll S, Sotlar K, George TI, Horny HP, Valent P, Reiter A, Kluin-Nelemans HC. Midostaurin improves quality of life and mediator-related symptoms in advanced systemic mastocytosis. J Allergy Clin Immunol. 2020 Aug;146(2):356-366.e4. doi: 10.1016/j.jaci.2020.03.044. Epub 2020 May 11. PMID 32437738
- [Derived] Gotlib J, Kluin-Nelemans HC, George TI, Akin C, Sotlar K, Hermine O, Awan FT, Hexner E, Mauro MJ, Sternberg DW, Villeneuve M, Huntsman Labed A, Stanek EJ, Hartmann K, Horny HP, Valent P, Reiter A. Efficacy and Safety of Midostaurin in Advanced Systemic Mastocytosis. N Engl J Med. 2016 Jun 30;374(26):2530-41. doi: 10.1056/NEJMoa1513098. PMID 27355533

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 29 centers in 12 countries worldwide (Australia, Austria, Belgium, Canada, France, Germany, Netherlands, Norway, Poland, Turkey, United Kingdom, United States).
Pre-assignment Details: The Participant Flow was on the Full Analysis Set (FAS), the Baseline Characteristics were done on the FAS and Primary Efficacy Population (PEP). The Efficacy analysis was done on the PEP (except for the Overall Survival which was done on FAS and PEP). The Safety analysis was done on the Safety Set (SS).
Period: Overall Study
Arm/Group | Midostaurin (PKC412)
Started (All patients to whom study treatment had been assigned (FAS)) | 116
Safety Set (SS) (All patients who received at least one dose of study drug) | 116
Primary Efficacy Population (PEP) (FAS patients meeting diagnostic criteria for ASM/MCL presenting at least one measurable C-finding) | 89
Completed | 0
Not Completed | 116
Not completed — Adverse Event | 35
Not completed — Subject withdrew consent | 11
Not completed — Lost to Follow-up | 2
Not completed — Administrative problems | 14
Not completed — Death | 9
Not completed — Disease progression | 43
Not completed — Protocol deviation | 2

BASELINE CHARACTERISTICS:
Population: The Participant Flow was on the Full Analysis Set (FAS), the Baseline Characteristics were done on the FAS and Primary Efficacy Population (PEP). The Efficacy analysis was done on the PEP (except for the Overall Survival which was done on FAS and PEP). The Safety analysis was done on the Safety Set (SS).
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 111
  More than one race | 0
  Unknown or Not Reported | 3
Age Continuous (PEP) [Mean (Standard Deviation); unit: Years] — Population: Primary Efficacy Population (PEP)
  Years
    number analyzed (Participants) | 89
    (all) | 63.0 (11.59)
Sex: Female, Male (PEP) [Number; unit: Participants] — Population: Primary Efficacy Population (PEP)
  Participants
    PEP (n=89) - Female: number analyzed (Participants) | 89
    PEP (n=89) - Female | 32
    PEP (n=89) - Male: number analyzed (Participants) | 89
    PEP (n=89) - Male | 57
Race (PEP) [Number; unit: Participants] — Population: Primary Efficacy Population (PEP)
  Participants
    PEP (n=89) - Black: number analyzed (Participants) | 89
    PEP (n=89) - Black | 1
    PEP (n=89) - White: number analyzed (Participants) | 89
    PEP (n=89) - White | 86
    PEP (n=89) - Other/Missing: number analyzed (Participants) | 89
    PEP (n=89) - Other/Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the percentage of participants who classified as confirmed responders (Major Response (MR) or Partial Response (PR)) by the adjudication of the SSC and based on a Modified Valent Criteria.
  A major responder had complete resolution of at least one C-Finding and no progression in other C-Findings. A partial responder showed a measurable improvement in one or more C-Finding(s) without confirmed progression in other C-Findings. A C-Finding was a Clinical Finding, which was considered by the investigator and corroborated by the Study Steering Committee (SSC) Chairperson or designee, attributable to the mast cell disease component and not the associated hematological clonal non-mast cell lineage disease (AHNMD) component or any other cause.
Time Frame: 6 months
Population: Primary Efficacy Population: participants assigned to study treatment who met diagnostic criteria for aggressive systemic mastocytosis or mast cell leukemia and presented with at least 1 measurable C-Finding at study entry and/or participants with transfusion dependent anemia due to their underlying disease at study entry as confirmed by the SCC.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 89
Percentage of participants | 59.6 [48.6 to 69.8]
Statistical Analysis 1: Comparison: Midostaurin (PKC412); Test type: Other — Single arm study; p < 0.001, Exact Binomial Test — Null hypothesis: ORR <= 30% Alternative hypothesis: ORR >= 50%; Exact Binomial 95% Confidence Interval

2. Secondary Outcome: Median Time to Duration of Response (DoR)
Description: The Duration of response (DoR) was defined as the time from first onset of confirmed response (MR or PR) to the date of first documented and confirmed progression or death due to ASM/MCL.
Time Frame: Up 5 years
Population: Primary Efficacy Population (PEP), which consisted of all participants with a confirmed response, was considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 89
Months | 31.4 [10.8 to NA] — Not Estimable because no event occured after median survival time

3. Secondary Outcome: Median Time to Response (TTR)
Description: The Time to response (TTR) was defined as the time from start of treatment until the date of onset of confirmed response (MR or PR).
Time Frame: Up 5 years
Population: Primary Efficacy Population (PEP), which consisted of all participants with a confirmed response, was considered.
Measure: Median (Full Range); unit: Months
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 89
Months | 0.3 [0.1 to 3.7]

4. Secondary Outcome: Median Time to Progression-Free Survival (PFS)
Description: The Progression-free survival (PFS) is defined as the time from start of treatment to the date of the first documented and confirmed progression or death due to any cause.
Time Frame: Up 5 years
Population: Primary Efficacy Population (PEP), which consisted of all participants with a confirmed response, was considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 89
Months | 17.0 [10.2 to 24.8]

5. Secondary Outcome: Median Time to Overall Survival (OS)
Description: The Overall Survival (OS) is defined as the time from start of treatment to the date of death due to any cause.
Time Frame: Up 5 years
Population: Primary Efficacy Population (PEP), which consisted of all participants with a confirmed response and the Full Analysis Set (FAS), which consisted of all patients who received at least one dose of study drug were considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 116
Months
  Primary Efficacy Population (PEP) (n=89): number analyzed (Participants) | 89
  Primary Efficacy Population (PEP) (n=89) | 26.8 [17.6 to 34.4]
  Full Analysis Set (FAS) (n=116) | 28.7 [20.3 to 38.0]

6. Secondary Outcome: Long-term Safety and Tolerability of Midostaurin
Description: Analysis of frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC)
Time Frame: Up to 30 days after last dose of study treatment
Population: Safety Set (SS)
Measure: Number; unit: Percentage of participants
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 116
Percentage of participants
  AEs by Primary System Organ Class (SOC) (n=116) | 100
  SAEs by Primary System Organ Class (SOC) (n=88): number analyzed (Participants) | 88
  SAEs by Primary System Organ Class (SOC) (n=88) | 75.9
  Deaths by Primary System Organ Class (SOC) (n=25): number analyzed (Participants) | 25
  Deaths by Primary System Organ Class (SOC) (n=25) | 21.6

7. Secondary Outcome: Histopathologic Response
Description: Histopathologic response was summarized to demonstrate the change from baseline in percentage of mast cell infiltrations in the Bone Marrow (BM) and related serum tryptase levels.
Time Frame: Up 5 years
Population: Primary Efficacy Population (PEP); for each patient, the best improvement relative to Baseline was considered.
Measure: Number; unit: Percentage of participants
Arm/Group | Midostaurin (PKC412)
Number analyzed (Participants) | 89
Percentage of participants
  >50% decrease in mast cell (MC) (n=41): number analyzed (Participants) | 41
  >50% decrease in mast cell (MC) (n=41) | 46.1
  >0-<=50% decrease in mast cell (MC) (n=19): number analyzed (Participants) | 19
  >0-<=50% decrease in mast cell (MC) (n=19) | 21.3
  >50% decrease in serum tryptase (n=52): number analyzed (Participants) | 52
  >50% decrease in serum tryptase (n=52) | 58.4
  >0-<=50% decrease in serum tryptase (n=25): number analyzed (Participants) | 25
  >0-<=50% decrease in serum tryptase (n=25) | 28.1

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 8 years and 7 months.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious adverse events fields "number of deaths resulting from adverse events" all those deaths, resulting from serious adverse events that are deemed to be causally related to treatment by the investigator.
Arm/Group | Midostaurin (PKC412)
All-Cause Mortality (participants affected / at risk) | 25/116
Serious Adverse Events (participants affected / at risk) | 88/116
Other Adverse Events (participants affected / at risk) | 115/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midostaurin (PKC412) (N=116)
Anaemia (Blood and lymphatic system disorders) | 8
Coagulopathy (Blood and lymphatic system disorders) | 1
Cytopenia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Granulocytopenia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Mastocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Splenic infarction (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Extrasystoles (Cardiac disorders) | 1
Heart valve incompetence (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Right ventricular failure (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Aplasia (Congenital, familial and genetic disorders) | 1
Ear disorder (Ear and labyrinth disorders) | 1
Papilloedema (Eye disorders) | 1
Retinopathy hypertensive (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 5
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Gastric varices haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal mass (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Varices oesophageal (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 3
General physical health deterioration (General disorders) | 2
Generalised oedema (General disorders) | 1
Malaise (General disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 3
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 7
Bile duct stenosis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Campylobacter colitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Malaria (Infections and infestations) | 1
Nocardiosis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 11
Sepsis (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Splenic infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Wound infection (Infections and infestations) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Transfusion related complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 1
Bleeding time prolonged (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Electrocardiogram ST segment depression (Investigations) | 1
Troponin increased (Investigations) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haematological malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Calculus urinary (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 5
Renal impairment (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 3
Heart valve operation (Surgical and medical procedures) | 1
Arterial occlusive disease (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haemodynamic instability (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Peripheral artery stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midostaurin (PKC412) (N=116)
Anaemia (Blood and lymphatic system disorders) | 39
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 23
Vertigo (Ear and labyrinth disorders) | 6
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 34
Abdominal pain upper (Gastrointestinal disorders) | 10
Ascites (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 62
Dyspepsia (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 94
Vomiting (Gastrointestinal disorders) | 77
Chills (General disorders) | 6
Fatigue (General disorders) | 33
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 41
Pain (General disorders) | 7
Pyrexia (General disorders) | 30
Bronchitis (Infections and infestations) | 8
Cystitis (Infections and infestations) | 7
Oral herpes (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 14
Viral upper respiratory tract infection (Infections and infestations) | 20
Contusion (Injury, poisoning and procedural complications) | 7
Alanine aminotransferase increased (Investigations) | 6
Amylase increased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 9
Blood creatinine increased (Investigations) | 6
Electrocardiogram QT prolonged (Investigations) | 12
Gamma-glutamyltransferase increased (Investigations) | 11
Lipase increased (Investigations) | 11
Weight decreased (Investigations) | 10
Decreased appetite (Metabolism and nutrition disorders) | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 24
Back pain (Musculoskeletal and connective tissue disorders) | 26
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Disturbance in attention (Nervous system disorders) | 8
Dizziness (Nervous system disorders) | 16
Headache (Nervous system disorders) | 29
Paraesthesia (Nervous system disorders) | 6
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 13
Insomnia (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 24
Rash (Skin and subcutaneous tissue disorders) | 7
Flushing (Vascular disorders) | 8
Haematoma (Vascular disorders) | 6
Hypotension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.